CLINICAL TRIAL: NCT05001958
Title: Understanding the Mechanisms of Action Observation as a Rehabilitation Intervention for Stroke
Brief Title: Action Observation as a Rehabilitation Intervention for Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Georgia Institute of Technology (Other)
Responsible Party: Principal Investigator, Veronica Thessing Rowe, Assistant Professor, Georgia State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H21185-GT
Record Dates: First submitted 2021-08-03; First posted 2021-08-12 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Action observation (Experimental)
  Interventions: Behavioral: Action observation

INTERVENTIONS:
Behavioral: Action observation — Participants will view a video of a task performed by a non-disabled actor and then the participants perform the task from the video with their weaker arm & hand.

SUMMARY:
One way to help a stroke survivor learn how to use their arm and hand again is to have them watch and replicate "normal" arm and hand movements. This type of intervention is called action observation (AO) and has emerged as a potentially powerful therapeutic tool to improve stroke rehabilitation for the weakened arm and hand. AO involves the patient's visual observation of video recorded intact body movements with the intent to perform the same task with their weakened arm and hand. There is behavioral evidence in stroke survivors that movement skills usually gained through physical practice can also be acquired through observation of the skill alone. In preliminary research performed in Dr. Lewis Wheaton's lab at Georgia Tech, AO has been successfully implemented for persons with arm and hand amputations learning how to use their prostheses. AO training in patients with amputations revealed that their movement is improved when they focus their eye gaze on specific aspects of the movement in the video that may maximally benefit the patient. It is unknown if these eye gaze patterns may serve as the mechanism behind AO and differ among those with mild or moderate movement impairments due to stroke. In this study, the investigators seek to identify if experience with AO in stroke survivors with varying levels of impairment has a similar emergence of eye gaze patterns found in people with amputations. The investigators hypothesize that AO augments visuomotor strategies to help support improved movement and enhance rehabilitation strategies in stroke survivors with mild and moderate impairments. The goal of this work is to utilize eye gaze tracking approaches to understand this phenomenon. In addition, the investigators will identify the feasibility of implementing and assessing AO on eye gaze in stroke survivors.

DETAILED DESCRIPTION:
Arm and hand impairments after stroke significantly limit daily activities and negatively impact quality of life. Action observation (AO) has emerged as a potentially powerful therapeutic intervention to improve stroke rehabilitation for the weakened arm and hand. AO involves the patient's visual observation of video recorded intact body movements from a non-disabled actor with the intent to perform the same skill task. There is behavioral evidence in stroke survivors that movement skills usually acquired through physical practice can also be acquired through observation of the movement skill alone. In preliminary research performed in Dr. Lewis Wheaton's lab at Georgia Tech, AO has been successfully implemented for persons with arm and hand amputations learning how to use their prostheses. Where the patient focuses their eye gaze on the video being observed has been shown to be key in improving their movement. That is, improved movement is associated with specific eye gaze patterns focused movement strategies observed in the non-disabled actor. It is unknown if these mechanisms of eye gaze patterns are also exhibited in stroke survivors, or if they are differentiated between those with varying levels of movement impairment. In this study, the investigators seek to identify if experience with AO in stroke survivors influences a similar emergence of gaze patterns found in people with amputations. In addition, the investigators seek to explore the differences in eye gaze and movement in stroke survivors who exhibit either mild or moderate impairments. The expected outcome of finding eye gaze strategy patterns that are most beneficial in improving movement of the arm and hand after stroke can enhance the implementation of AO by instructing participants with guided cuing to focus on specific areas of interest in the videos.

Twenty participants with either mild or moderate weakness in their arm and hand due to stroke will complete the AO intervention with eye gaze and movement assessments. The goal of this work is to implement eye-tracking approaches to understand how AO augments visuomotor strategies (i.e., the mechanism) to help improve movement and enhance rehabilitation strategies in stroke survivors with varying levels of impairments.

Aim 1: Evaluate how AO influences eye gaze strategies in stroke survivors as a function of stroke severity. Hypothesis: There are eye gaze pattern strategies in stroke survivors that differ between those with mild and moderate movement impairments. Eye gaze pattern strategies will be assessed during AO, i.e., while watching the videos between participants that are mildly and moderately impaired.

Aim 2: Evaluate the relationship between eye gaze strategies and arm and hand movement in stroke survivors as a function of stroke severity. Hypothesis: AO influences the relationship of arm and hand movement with varying gaze pattern strategies in stroke survivors with mild or moderate movement impairments. Arm and hand functional movement will be assessed following AO between participants that are mildly and moderately impaired.

Aim 3: Identify the feasibility of implementing and assessing AO in stroke survivors. Hypothesis: There are specific factors that facilitate or hinder the recruitment, retention, and completion of this protocol. Feasibility of this protocol will be assessed to provide guidance for future research efforts in the stroke population.

ELIGIBILITY:
Inclusion Criteria:

* stroke experienced at 18 years of age or older
* not undergoing any physical rehabilitation during the time enrolled in this study
* mild to moderate impairments in the more affected arm and hand (i.e., movement and coordination scores on the Fugl-Meyer Assessment between 20 and 55)
* no cognitive impairments (mini-mental state examination ≥ 24/30)
* normal or corrected vision (National Institutes of Health Stroke Scale = 0)

Exclusion Criteria:

* any uncorrected impairment to the visual field, such as spatial neglect or inattention (i.e., decreased awareness/perception of objects or people in a section of the visual field) (National Institutes of Health Stroke Scale > 1)
* inability to communicate and participate effectively for assessments and intervention sessions (mini-mental state examination and National Institutes of Health Stroke Scale) upper arm and hand movement impairment that is severe (Fugl-Meyer Assessment < 20) or non-existent (Fugl-Meyer Assessment > 55)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Eye gaze pattern | Eye gaze recorded in one day during the 3 blocks of video watching (action observation)
  Eye gaze patterns will be collected with a Pupil Labs Eye Camera (Berlin, Germany; 200 Hz, binocular) throughout the experiment. The participants will don eye tracking glasses that feature two pupil cameras which track the participants' pupils relative to the world, which records what participants see in their line of vision. Eye gaze will identify areas of interest of the SRTT (movement task).
Arm and hand movement with the Serial Reaction Time Test (SRTT) | Arm and hand movement recorded in one day during the 3 blocks of physical performance of the SRTT
  The participants' arm and hand movement will be analyzed when the participants perform the SRTT action using a Sensor Ascension trakSTAR system (Motion Monitor, Chicago). Electromagnetic sensors (MotionMonitor, Chicago) will be placed at key locations on the participant's arm and hand that they are using to complete the SRTT.

CONTACTS AND LOCATIONS:
Overall Officials: Veronica T Rowe, PhD, OTR/L, Principal Investigator — Georgia State University
Locations (1):
- Georgia Tech, Atlanta, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No